CLINICAL TRIAL: NCT06547424
Title: A Randomized, Controlled, Double-Blind Phase I Clinical Study of Chondroitin Sulfate Supplementation for Treatment of Necrotizing Enterocolitis
Brief Title: Phase I Clinical Study of Chondroitin Sulfate for Treatment of NEC
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Project plan was abandoned.
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Troy Markel, Professor of Surgery, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 23893
Record Dates: First submitted 2024-08-07; First posted 2024-08-09 (Actual); Last update posted 2025-10-10 (Actual); Status verified 2025-10

CONDITIONS: Necrotizing Enterocolitis; Intestinal Ischemia
Keywords: chondroitin sulfate
MeSH Terms: conditions — Enterocolitis, Necrotizing | interventions — Chondroitin Sulfates

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Chondroitin sulfate (Experimental): Neonates with Bell's Stage 2 NEC will receive chondroitin sulfate (20mg/kg/day) dissolved in 1-2 mil of milk or formula for 2 days
  Interventions: Drug: Chondroitin sulfate
- Placebo (Placebo Comparator): Neonates with Bell's Stage 2 NEC will receive 1-2 ml of milk or formula placebo for 2 days
  Interventions: Drug: Chondroitin sulfate

INTERVENTIONS:
Drug: Chondroitin sulfate — Neonates with Bell's Stage 2 NEC will be given chondroitin sulfate (20mg/kg/day) mixed with 1-2 ml of milk or formula for 2 days

SUMMARY:
The goal of this phase 1 double blind, randomized controlled trial is to determine the safety of chondroitin sulfate supplementation in the neonates with necrotizing enterocolitis. The main questions the study aims to answer are:

Is chondroitin sulfate safe to administer in the neonatal NEC population, and will it have a beneficial profile in the short term intestinal and long term neurodevelopmental sequelae of NEC? Researchers will compare all cause mortality, progression to surgery, systemic inflammatory markers, and long term neurodevelopmental outcomes in those NEC patients who receive chondroitin sulfate compared to those who receive milk or formula placebo.

DETAILED DESCRIPTION:
Necrotizing Enterocolitis (NEC) is a devastating intra-abdominal emergency that primarily affects premature infants and is characterized by abdominal distention, extreme illness, and intestinal necrosis-with mortality rates that range from 20-30%. Despite earnest research, there have been no significant advances in our ability to treat this disease within the last several decades, making NEC an unmet medical need.

Neurodevelopmental impairment (NDI) is a detrimental sequela in infants with NEC and carries an incidence of approximately 40%. NDI is believed to be a result of the systemic inflammatory response and pathogenic signaling cascades associated with NEC, resulting in white-matter injury, alterations in brain parenchyma, and loss of brain matter volume-which then manifest in later life as cognitive and motor deficits, autism, and cerebral palsy. Novel therapeutic strategies to treat or prevent NEC and its long-term sequelae would have a significant impact on reducing morbidity and mortality in this fragile population.

Our long-term goal is to develop effective methods for the prevention and treatment of NEC and its neurodevelopmental sequelae. In this regard, the use of human breast milk (HM) is an important preventative strategy to reduce the incidence of NEC. In one study, 7.2% of infants receiving formula developed NEC while only 1.2% of infants exclusively being fed breastmilk developed NEC. This would suggest that protective compounds exist in human breastmilk that may prevent NEC. However, despite the beneficial properties of human breastmilk, it's important to note that breast milk has not been shown to eliminate NEC. Therefore, finding protective compounds in HM that could be utilized as a formula additive or breast milk booster would be highly effective in further preventing and treating NEC. A prominent glycosoaminoglycan gaining clinical interest is chondroitin sulfate (CS), which comprises over half of the normal GAG content in HM and is surprisingly nonexistent in most major infant formulas. Additionally, the concentration of CS in HM is higher in preterm mothers than in term mothers, thereby suggesting some evolutionary importance for this compound to preterm infants6.

A review of the prior rigor of research suggests that CS decreases blood lipopolysaccharide (LPS) levels in mice experiencing stress, reduces invasion and translocation of bacteria within the intestine, restores repressed fecal short-chain fatty acids, and alters the intestinal microbiome. We have appreciated beneficial effects of CS in protecting the intestine during experimental NEC. A possible mechanism of action surrounds its modulation of the Th17 immune cell profile. An increase in Th17 cells and intestinal NFĸΒ phosphorylation has long been recognized as contributing molecular factors in NEC. Furthermore, IL-17 is an important effector cytokine of Th17 cells and is involved in the pathogenesis of acute neuroinflammatory conditions.

The overarching goal of this project is to perform a randomized, controlled, double blind phase 1 clinical trial to assess the short- and long-term safety profiles of chondroitin sulfate for the treatment of necrotizing enterocolitis in the neonatal population. Preliminary data from murine and porcine animal models in our lab have shown protection against the intestinal and neurodevelopmental sequelae of NEC. CS has previously been considered a food supplement and therefore is not regulated by the FDA. It has been classified as Generally Recognized as Safe by the FDA and has been used in adult clinical trials without increased safety concerns. We therefore hypothesize that CS will be safe to administer in the neonatal NEC population and will have a beneficial safety profile in the short term intestinal and long term neurodevelopmental sequela of NEC. To test these hypotheses, we propose the following Specific Aims:

1. Assess the short-term safety profile of CS supplementation in the neonatal NEC population and its impact on mortality, progression to surgery, and the systemic inflammatory profile. Adverse events, progression to surgery, and all-cause mortality will be assessed in preterm low birth weight infants with Bell's Stage II NEC. Additionally, the ability of CS to modulate the immune cell profile and systemic inflammatory response will be assessed.
2. Determine the impact of chondroitin sulfate supplementation on neurodevelopmental outcomes in the NEC population as a marker of long-term safety. To assess long-term safety, neurodevelopmental impairment of infants receiving CS will be compared to placebo at both 1- and 2-years following administration. We hypothesize that CS infants would have similar, if not improved NDI compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

1. NICU patient at Riley Hospital for Children
2. Weight of less than 2500g at time of NEC diagnosis
3. Patient must have a diagnosis of Bell's Stage 2 necrotizing enterocolitis

Exclusion Criteria:

1. Severe cardiac or neurological congenital anomalies
2. Previous history of NEC
3. History of abdominal surgery or other intestinal congenital anomalies
4. Renal failure or renal impairment necessitating dialysis
5. Any end-stage organ disease, infection, or condition, which in the opinion of the Investigator, makes the patient an unsuitable candidate for treatment
6. Receipt of another investigational therapy
7. Informed consent is unable to be obtained from parent or legally authorized representative
8. Patient is a ward of the court system

Ages: 1 Hour to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2025-01 (Estimated); Primary Completion 2028-12 (Estimated); Study Completion 2029-03 (Estimated)

PRIMARY OUTCOMES:
Mortality | 14 and 28 days post intervention
Progression to need for surgery | 14 and 28 days post intervention
  Infants with Stage 2 NEC can progress to stage 3 NEC and require surgery to remove intestinal tissue. This rate will be compared in the intervention and placebo arms

SECONDARY OUTCOMES:
Systemic inflammatory markers | 14 and 28 days post intervention
  Blood will be assessed for common inflammatory markers
Neurodevelopmental impairment (NDI) | 1 and 2 years post intervention
  NDI will be assessed at 1 and 2 years post intervention. eurodevelopmental impairment will be defined as any of the following: moderate to severe cerebral palsy (CP) with Gross Motor Function Classification System level ≥ 2, Bayley-IV cognitive composite score <85, severe bilateral visual impairment consistent with vision <20/200, or permanent hearing loss despite amplification that prevents communication or understanding the examiner

CONTACTS AND LOCATIONS:
Locations (1):
- Riley Hospital for Children, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
Results of the study will be published at completion
Supporting Information: Study Protocol, CSR
Time Frame: within 6 months of study completion